CLINICAL TRIAL: NCT06707649
Title: The Effectiveness of Self-Management Education and Telephone Follow-up on Self-Care Agency and Symptom Management in Patients with COPD Exacerbation: a Randomized Controlled Study
Brief Title: The Effectiveness of Self-Management Education and Telephone Follow-up in Patient with COPD Exacerbation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Yasemin CEYHAN, Assistant Proffesor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/03/43
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-09

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Symptom Management; Self-care Agency
Keywords: COPD (Chronic Obstructive Pulmonary Disease); Symptom Management; Telephone Follow-up; Self-care Agency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Education+Telephone Follow-up (Experimental): Patients in this group will receive self-management education during the 3 days when they are in the hospital. On the first day of the training, COPD disease, causes of the disease, symptoms, reasons for alleviating complaints, practical information for living comfortably with COPD will be given. On the second day, emergency situations in COPD, what is an exacerbation and prevention suggestions and diaphragmatic breathing-cough exercises will be taught. On the last day, training will be given on pursed lip breathing, medication use, oxygen and nebulizer treatments. Patients will receive their first call one week after discharge. The calls will be scheduled weekly during the first month, biweekly in the second month, and monthly starting from the third month. During the calls, it is planned to repeat the educational content and answer the patient's questions. All scales are planned to be re-administered at 1, 3, and 6 months.
  Interventions: Other: Self Management Education; Other: Telephone Follow-up
- Education (Experimental): Patients in this group will receive self-management education during the 3 days when they are in the hospital. On the first day of the training, COPD disease, causes of the disease, symptoms, reasons for alleviating complaints, practical information for living comfortably with COPD will be given. On the second day, emergency situations in COPD, what is an exacerbation and prevention suggestions and diaphragmatic breathing-cough exercises will be taught. On the last day, training will be given on puckered lip breathing, medication use, oxygen and nebulizer treatments. Patients in this group will not receive telephone follow-up. All scales are planned to be re-administered at 1, 3, and 6 months.
  Interventions: Other: Self Management Education
- Standard Care (Active Comparator): Patients in this group will receive standard care. Education and telephone follow-up will not be applied. All scales are planned to be re-administered at 1, 3, and 6 months.
  Interventions: Other: Self Management Education; Other: Telephone Follow-up

INTERVENTIONS:
Other: Self Management Education — Patients in this group will receive self-management education during the 3 days when they are in the hospital. On the first day of the training, COPD disease, causes of the disease, symptoms, reasons for alleviating complaints, practical information for living comfortably with COPD will be given. On the second day, emergency situations in COPD, what is an exacerbation and prevention suggestions and diaphragmatic breathing-cough exercises will be taught. On the last day, training will be given on pursed lip breathing, medication use, oxygen and nebulizer treatments. The education will be accompanied by a educational booklet prepared by researchers and expert opinion.
Other: Telephone Follow-up — Patients will receive their first call one week after discharge. The calls will be scheduled weekly during the first month, biweekly in the second month, and monthly starting from the third month. During the calls, it is planned to repeat the educational content and answer the patient's questions.
  Arms: Education+Telephone Follow-up; Standard Care

SUMMARY:
According to the 2024 GOLD guidelines, Chronic Obstructive Pulmonary Disease (COPD) is defined as heterogeneous lung condition characterized by chronic respiratory symptoms (dyspnea, cough, sputum production, and/or exacerbations) due to abnormalities of the airways (bronchitis, bronchiolitis) and/or alveoli (emphysema) that cause persistent, often progressive, airflow obstruction. COPD is one of the leading causes of mortality and morbidity in Turkey and worldwide. Since COPD is an incurable and lifelong disease, it is important for patients to have high levels of self-management.

The main questions it aims to answer are:

1. Does self-management education and telephone follow-up intervention effect self-care agency and symptom management in people with COPD exacerbation?
2. Does self-management education effect self-care agency and symptom management in people with COPD exacerbation? This study will evaluate the effect of self-management education and telephone follow-up on self-care agency and symptom management. Patients hospitalized with COPD exacerbation will be trained in the hospital and will be followed up by phone call after discharge. During the study, 3 groups were planned; Group 1 will be educated and followed up by telephone Group 2 will only receive education and no telephone follow-up. Group 3 will not receive education and telephone follow-up, only standard care. It is planned to collect the data from the patients at the beginning of the study, at 1, 3 and 6 months.

Main outcomes:

* Level of self-care agency
* Level of symptom management The results obtained will be interpreted by comparing between 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD for the last 1 year
* Diagnosis of Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage III or IV COPD documented by pulmonary function testing
* Patients hospitalized for acute exacerbation of COPD;
* Hospitalized for at least 3 days
* Having a personal mobile phone and the ability to use it,
* Being enough conscious and oriented to answer the questions,
* Voluntary patients

Exclusion Criteria:

* Under 18 years old
* Withdrawal from the study at any phase
* Inability to be contacted by phone/mobile phone,
* Patient death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
mMRC Dyspnea Scale | will be re-administered in the pre-test and interviews with patients at 1, 3 and 6 months
  It is used to rate the effects of breathlessness in daily activities. The scale was developed and modified by the British Medical Research Council (MRC) to determine the course of breathlessness in respiratory diseases. The MMRC is a five-item scale based on various movements that cause shortness of breath.
The COPD Assessment Test | will be re-administered in the pre-test and interviews with patients at 1, 3 and 6 months
  The Turkish reliability and validity of the scale, which consists of eight questions to assess health status in COPD, was conducted by Yorgancıoğlu et al. in 2012. The COPD Assessment Test provides assessment of conditions such as sputum, shortness of breath, cough, fatigue, and sleep. Each question is scored between 0 (no symptoms) and 5 (severe symptoms). The scores of the questions in the test are between "0-40". The higher the score, the more severe the disease and the worse the health status.
Clinical COPD Questionnaire (CCQ) | will be re-administered in the pre-test and interviews with patients at 1, 3 and 6 months
  It is a 10-item questionnaire (4 items for symptoms, 4 items for functional status and 2 items for mental status) that measures clinical control to assess functional status, mental status and symptoms and is valid and reliable in Turkish.
The Modified Borg Dyspnea Scale | will be re-administered in the pre-test and interviews with patients at 1, 3 and 6 months
  The Modified Borg Dyspnea Scale was developed by Borg in 1970 to measure the effort expended during exercise and the level of dyspnea felt at the maximum level at which exercise has to be stopped. The severity of dyspnea on the scale is expressed by ten items defined from "0 (none)" to "10 (very severe)". The severity of exertion during exercise is graded according to this scoring to determine the level of dyspnea.

SECONDARY OUTCOMES:
Self-Care Agency | will be re-administered in the pre-test and interviews with patients at 1, 3 and 6 months
  The scale was developed by Kearney and Fleicher (1979) in English with 43 items, and its Turkish validity and reliability was shortened to 35 items by Nursen Nahcivan (Nahcivan, 1994; Nahcivan 2004). The scale focuses on individuals self-assessment of their involvement in self-care activities. Each statement is scored from 0 to 4. Individuals orientation towards self-care is determined by participants responses on a 5-point Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin CEYHAN, PhD, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kirsehir Training and Research Hospital, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No